CLINICAL TRIAL: NCT03690999
Title: Impact of a Prebiotic Supplement on Microbiome, Immune System, and Metabolic Status of Older Adults
Brief Title: The RAMP Study - Rejuvenation of the Aging Microbiota With Prebiotics
Acronym: RAMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Justin L. Sonnenburg, Associate Professor of Microbiology and Immunology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 47252
Record Dates: First submitted 2018-09-17; First posted 2018-10-01 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Microbiome; Immune Function; Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo group (Placebo Comparator): Placebo product
  Interventions: Dietary Supplement: Placebo
- Prebiotic Supplement, low dose (Experimental)
  Interventions: Dietary Supplement: Prebiotic supplement
- Prebiotic Supplement, high dose (Experimental)
  Interventions: Dietary Supplement: Prebiotic supplement

INTERVENTIONS:
Dietary Supplement: Placebo — Placebo product
  Arms: Placebo group
Dietary Supplement: Prebiotic supplement — Prebiotic supplement
  Arms: Prebiotic Supplement, high dose; Prebiotic Supplement, low dose

SUMMARY:
An individual's immune and metabolic status is coupled to consumed carbohydrates. Complex carbohydrates that are not digested by human enzymes may influence host biology by impacting microbiota composition and function, or act in a yet-unknown microbiota-independent manner. Prebiotics offer a promising safe route to influence host health, possibly via the microbiota. However, it remains largely unknown to what extent immune function and metabolism can be modulated by prebiotics.

DETAILED DESCRIPTION:
The objective of this study is to define the impact of a prebiotic supplement on microbiome, immune system, and metabolic status in older adults. This study will determine the degree to which a prebiotic supplement can 1) regulate immune status and function including reducing chronic, systemic inflammation as assessed by high dimensional immune profiling, 2) alter microbiota composition and function, 3) impact the microbiota metabolites-potential normalizers of metabolic and immune dysfunction, and 4) alter metabolic markers.

ELIGIBILITY:
Inclusion Criteria:

* 60 years old and older
* Otherwise, healthy subjects willing and able to provide blood as well as stool specimens
* Must be able to provide signed and dated informed consent and be willing to follow protocol

Exclusion Criteria:

* Body Mass Index >= 40
* LDL-C > 190 mg/dL
* Systolic Blood Pressure >160 mmHg OR Diastolic Blood Pressure > 90 mmHg
* Use of any of the following drugs/supplements within the last 2 months:

  * systemic antibiotics, antifungals, antivirals or antiparasitics (intravenous, intramuscular, or oral);
  * corticosteroids (intravenous, intramuscular, oral, nasal or inhaled)
  * cytokines
  * methotrexate or immunosuppressive cytotoxic agents
  * metformin
  * proton pump inhibitors (PPIs)
* Regular use of any of the following medications:

  * regular dose aspirin (>81mg/day)
  * opiate pain medication
* Use of large doses of commercial probiotics consumed (greater than or equal to 10-8 cfu or organisms per day) - includes tablets, capsules, lozenges, chewing gum or powders in which probiotic is a primary component. Ordinary dietary components such as fermented beverages/milks, yogurts, foods do not apply.
* Acute disease at the time of enrollment. Acute disease is defined as the presence of a moderate or severe illness with or without fever. Examples include flu or gastroenteritis. Defer sampling until subject recover.
* Chronic, clinically significant, unstable (unresolved, requiring on-going changes to medical management or medication) pulmonary, cardiovascular, gastrointestinal, hepatic or renal functional abnormality, as determined by medical history. Type 2 diabetes, type 1 diabetes, and dialysis will be excluded.
* History of active uncontrolled gastrointestinal disorders or diseases including:

  * inflammatory bowel disease (IBD) including ulcerative colitis (mild-moderate-severe), Crohn's disease (mild-moderate-severe), or indeterminate colitis;
  * irritable bowel syndrome (IBS) (moderate-severe);
  * persistent, infectious gastroenteritis, colitis or gastritis, persistent or chronic diarrhea of unknown etiology, Clostridium difficile infection (recurrent) or Helicobacter pylori infection (untreated).
* History of active cancer in the past 3 years except for squamous or basal cell carcinomas of the skin that have been medically managed by local excision.
* Unstable dietary history as defined by major changes in diet during the previous month, where the subject has eliminated or significantly increased a major food group in the diet.
* Recent history of chronic excessive alcohol consumption defined as more than five 1.5-ounce servings of 80 proof distilled spirits, five 12-ounce servings of beer or five 5-ounce servings of wine per day; or > 14 drinks/week.
* Positive test for HIV, HBV or HCV.
* Any confirmed or suspected condition/state of immunosuppression or immunodeficiency (primary or acquired) including HIV infection.
* Surgery of the GI tract, with the exception of cholecystectomy and appendectomy, in the past five years. Any major bowel resection at any time.
* Regular/frequent use of smoking or chewing tobacco, e-cigarettes, cigars or other nicotine-containing products.
* Any confirmed or suspected autoimmune disease. Examples include multiple sclerosis and Graves disease.
* Veganism.
* Dairy allergies.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Immune status and function | Baseline and 6 weeks
  Change from baseline in Cytokine Response Score (CRS) at 6 weeks. The CRS is a single composite measure of cell-type specific activation of signaling pathways from ex vivo cytokine stimulation of blood samples. This provides a measure of immune response capacity which may be an indicator of immune fitness. The CRS will be calculated as described in Shen-Orr et al, Cell Systems, 2016. The CRS is the sum of 15 age-associated normalized cytokine responses identified in Shen-Orr et. al: In CD8+ T cells: IFNα pSTAT1, pSTAT3, pSTAT5; IL-6 pSTAT1, pSTAT3, pSTAT5; IFNγ pSTAT1; IL-21 pSTAT1; In CD4+ T cells: IFNα pSTAT5; IL-6 pSTAT5; In B cells: IFNα pSTAT1; in monocytes: IL-10 pSTAT3; IFNγ pSTAT3; IFNα pSTAT3; IL-6 pSTAT3. Each feature is calculated as the fold change of the protein in the stimulated condition relative to its level in the unstimulated condition. That value is then normalized to the feature's range: normalized = (x - xmin)/xmax. The 15 normalized values are summed for the CRS.

SECONDARY OUTCOMES:
Microbiota composition | Baseline and 6 weeks
  Change from baseline in alpha diversity at 6 weeks. We will be using number of observed sequence variants ("species") determined by standard 16S rRNA amplicon sequencing (V3-V5 region followed by DADA2 to define error-corrected sequence variants) as our primary metric of alpha diversity. Higher alpha diversity is better. The units are the # of sequence variants.
Microbiota function | Baseline and 6 weeks
  Change from baseline in composite of short-chain fatty acids (SCFA) concentration (ug/g stool: acetate + propionate + butyrate) at 6 weeks.
Weight | Baseline and 6 weeks
  Change from Baseline in weight at 6 weeks.
Waist Circumference | Baseline and 6 weeks
  Change from Baseline in waist circumference at 6 weeks.
Blood pressure | Baseline and 6 weeks
  Change from Baseline in blood pressure at 6 weeks.
Total Cholesterol | Baseline and 6 weeks
  Change from Baseline in total cholesterol at 6 weeks.
Triglycerides | Baseline and 6 weeks
  Change from Baseline in triglycerides at 6 weeks.
HDL-cholesterol | Baseline and 6 weeks
  Change from Baseline in HDL-cholesterol at 6 weeks.
Fasting Glucose | Baseline and 6 weeks
  Change from Baseline in fasting glucose at 6 weeks.
Fasting Insulin | Baseline and 6 weeks
  Change from Baseline in fasting insulin at 6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Justin Sonnenburg, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carter MM, Demis D, Perelman D, St Onge M, Petlura C, Cunanan K, Mathi K, Maecker HT, Chow JM, Robinson JL, Sabag-Daigle A, Sonnenburg ED, Buck RH, Gardner CD, Sonnenburg JL. A human milk oligosaccharide alters the microbiome, circulating hormones, and metabolites in a randomized controlled trial of older adults. Cell Rep Med. 2025 Aug 19;6(8):102256. doi: 10.1016/j.xcrm.2025.102256. Epub 2025 Jul 29. PMID 40738103
- See also: Study description — https://med.stanford.edu/nutrition/research/completed-studies/RAMPStudy.html

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-06-25): https://cdn.clinicaltrials.gov/large-docs/99/NCT03690999/SAP_000.pdf